CLINICAL TRIAL: NCT00704795
Title: Glucagon Responses Following Oral Glucose and Isoglycemic iv Glucose in Patients With Type 1 Diabetes - a Role for the Gastrointestinal Tract in Diabetic Hyperglucagonemia?
Brief Title: Glucagon Responses During Oral- and iv Glucose in Patients With Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Kristine Juul Hare/MD, Gentofte University Hospital, Copenhagen
Other Study IDs: H-D-2008-037
Record Dates: First submitted 2008-06-24; First posted 2008-06-25 (Estimated); Last update posted 2008-06-26 (Estimated); Status verified 2008-06

CONDITIONS: Hyperglucagonemia; Hyperglycemia; Diabetes Mellitus
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with type 1 diabetes mellitus
  Interventions: Other: Oral glucose tolerance test; Other: Isoglycemic iv glucose infusion
- 2: Healthy control subjects matched for body mass index (BMI), age and gender.
  Interventions: Other: Oral glucose tolerance test; Other: Isoglycemic iv glucose infusion

INTERVENTIONS:
Other: Oral glucose tolerance test — 50 g of waterfree glucose dissolved in 300 ml water is ingested over 5 minutes following a 10-h fast including liquids and medication (if any).
  Other Names: OGTT; 50 g-OGTT
Other: Isoglycemic iv glucose infusion — The plasma glucose curve obtained during a 50 g-OGTT (performed on a separate day) is copied using an adjustable iv glucose infusion (20% w/v) performed following a 10-h fast including liquids and medication (if any). The iv catheter is inserted into a peripheral vein in the hand/forearm.
  Other Names: Isoglycemic IVGTT

SUMMARY:
In order to evaluate the potential role of the gastrointestinal (GI) tract in the postprandial hyperglucagonemia, which characterizes type 1 diabetes mellitus (T1DM) (as well as type 2 diabetes mellitus (T2DM)), we wish to investigate the secretion of glucagon in patients with T1DM without residual beta-cell function during 50-g oral glucose tolerance test (OGTT) and during isoglycemic iv glucose infusion. By evaluating C-peptide negative patients with T1DM we aim to describe the glucagon response to glucose (+/-stimulation of the GI tract) independently of the potentially very important regulation of glucagon secretion by endogenous insulin secretion. A more detailed understanding of the inappropriate glucagon secretion in T1DM is highly needed in order to establish new intervention strategies in the future treatment of the growing numbers of T1DM patients.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian over 18 years with T1DM (diagnosed according to WHO's criteria) treated with long-acting insulin
* No residual beta-cell function (arginine test without increment in plasma C-peptide - see below)
* BMI <30 kg/m2
* Normal haemoglobin
* Informed consent

Exclusion Criteria:

* Residual beta-cell function (increment in plasma C-peptide during arginine test - see below)
* Known liver disease or affected liver enzymes (ALAT/ASAT > 2 x upper normal limit)
* Diabetic nephropathy (se-creatinin > 130 µM and/or albuminuria)
* Proliferative diabetic retinopathy (anamnestic)
* Treatment with medication that cannot be discontinued for 14 hours

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with type 1 diabetes mellitus and no residual beta-cell function (C-peptide negative)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Glucagon responses (as assessed by area under curve (AUC)) during 50-g oral glucose tolerance test (OGTT) and isoglycemic iv glucose infusion, respectively. | months

SECONDARY OUTCOMES:
Responses of glucagon-like peptide-1 (GLP-1), glucagon-like peptide-2 (GLP-2) and glucose-dependent insulinotropic polypeptide (GIP) as assessed by AUC during 50-g OGTT and isoglycemic iv glucose infusion, respectively. | months
GI-mediated glucose tolerance as assessed by the amount of glucose ingested as compared to the amount of glucose needed to mimic the OGTT curve during the iv glucose infusion. | Months

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD PhD, Principal Investigator — University Hospital, Gentofte, Copenhagen
Locations (1):
- Gentofte University Hospital, Hellerup, Hellerup, Denmark